CLINICAL TRIAL: NCT02426086
Title: A Randomized, Single-Blind, Multicenter Phase 2 Study to Evaluate the Activity of 2 Dose Levels of Imetelstat in Subjects With Intermediate-2 or High-Risk Myelofibrosis (MF) Relapsed/Refractory to Janus Kinase (JAK) Inhibitor
Brief Title: Study to Evaluate Activity of 2 Dose Levels of Imetelstat in Participants With Intermediate-2 or High-Risk Myelofibrosis (MF) Previously Treated With Janus Kinase (JAK) Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR107170; 63935937MYF2001 (Other: Geron Corporation); 2015-000946-41 (EudraCT Number)
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Imetelstat; GRN163L; Relapsed/refractory to JAKi; IMbark
MeSH Terms: conditions — Primary Myelofibrosis; Recurrence | interventions — imetelstat

STUDY DESIGN:
Who Masked: Participant
Masking Description: Initially single-blind; treatments unmasked after 1st Interim Analysis and continued as open-label treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Imetelstat 4.7 mg/kg (Experimental)
  Interventions: Drug: Imetelstat 4.7 mg/kg
- Imetelstat 9.4 mg/kg (Experimental)
  Interventions: Drug: Imetelstat 9.4 mg/kg

INTERVENTIONS:
Drug: Imetelstat 4.7 mg/kg — Participants received imetelstat 4.7 mg/kg of body weight as intravenous infusion on Day 1 of each 21-day cycle. Study drug was administered intravenously until disease progression, unacceptable toxicity, or study end.
  Arms: Imetelstat 4.7 mg/kg
Drug: Imetelstat 9.4 mg/kg — Participants received imetelstat 9.4 mg/kg of body weight as intravenous infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or study end.
  Arms: Imetelstat 9.4 mg/kg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 dose regimens of imetelstat in participants with intermediate-2 or high-risk myelofibrosis (MF) whose disease is relapsed after or is refractory to Janus Kinase (JAK) inhibitor treatment. Key secondary endpoint includes overall survival.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), multicenter (more than one hospital, medical school team or medical clinic work on a medical research study) study of 2 dosing regimens (treatment arms) of single-agent imetelstat in participants with intermediate-2 or high risk myelofibrosis (MF) whose disease is relapsed after or refractory to Janus Kinase (JAK) inhibitor treatment. The main study consists of 3 parts: Screening Phase (21 days before randomization); Treatment Phase (from randomization until study drug discontinuation); and Follow up Phase (until death, lost to follow-up, withdrawal of consent or study end, whichever occurs first). Participants received imetelstat 9.4 milligram (mg)/kilogram (kg) intravenously (IV) for every 3 weeks until disease progression, unacceptable toxicity, or study end OR imetelstat 4.7 mg/kg IV for every 3 weeks until disease progression, unacceptable toxicity, or study end. Initially, all participants were blinded to the treatment. After the first interim analysis, treatment for all participants was unblinded and participants assigned to the imetelstat 4.7 mg/kg arm could continue with their same imetelstat dose or have it increased to 9.4 mg/kg at the investigator's discretion. The percentage of spleen response and symptom response were evaluated as co-primary endpoints. Following completion of the primary analysis, participants benefiting from study treatment could continue to receive imetelstat in Extension phase for up to 2 years or until loss of benefit or unacceptable toxicity. Participants who had already stopped study treatment could enter the Extension phase to continue follow up for safety via serious adverse event collection and for survival status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis (PMF) according to the revised WHO criteria; or post-essential thrombocythemia-myelofibrosis (PET-MF) or post-polycythemia vera-myelofibrosis (PPV-MF) according to the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria.
* Dynamic International Prognostic Scoring System (DIPSS) intermediate-2 or highrisk MF.
* Measurable splenomegaly prior to study entry as demonstrated by palpable spleen measuring ≥ 5 cm below the left costal margin OR spleen volume of ≥ 450 cm^3 measured by magnetic resonance imaging (MRI).
* Active symptoms of MF as demonstrated by a symptom score of at least 5 points (on a 0 to 10 scale) on at least one of the symptoms or a score of 3 or greater on at least 2 of the symptoms.
* Documented progressive disease during or after Janus kinase (JAK) inhibitor therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.

Exclusion Criteria:

* Peripheral blood blast count of ≥ 10% or bone marrow blast count of ≥ 10%.
* Prior treatment with imetelstat.
* Any chemotherapy or MF-directed therapy, investigational drug, hydroxyurea, immunomodulatory or immunosuppressive therapy, corticosteroids or JAK inhibitor therapy ≤14 days prior to randomization.
* Major surgery within 4 weeks prior to randomization.
* Active systemic hepatitis infection requiring treatment (carriers of hepatitis virus are permitted to enter the study), of any type or known acute or chronic liver disease including cirrhosis.
* Prior history of hematopoietic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2020-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Clinical Team, Study Director — Geron Corporation
Locations (72):
- United States (29):
  - Birmingham, Alabama
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - Stanford, California
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Buffalo, New York
  - Lake Success, New York
  - New York, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Watertown, South Dakota
  - Nashville, Tennessee
  - Dallas, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Belgium (4):
  - Antwerp
  - Bruges
  - Brussels
  - Leuven
- Canada (3):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Montreal, Quebec
- France (6):
  - Angers
  - Lille
  - Marseille
  - Paris
  - Pierre-Bénite
  - Toulouse
- Germany (10):
  - Aachen
  - Cologne
  - Dresden
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Heidelberg
  - Leipzig
  - Mannheim
  - Rostock
- Israel (6):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Ramat Gan
  - Tel Aviv
- Italy (2):
  - Bergamo
  - Bologna
- Seoul, South Korea
- Spain (5):
  - Barcelona
  - Las Palmas de Gran Canaria
  - Madrid
  - Salamanca
  - Valencia
- Taiwan (2):
  - Chiayi City
  - Taipei
- United Kingdom (4):
  - Birmingham
  - Glasgow
  - London
  - Oxford

REFERENCES:
- [Derived] Mascarenhas J, Komrokji RS, Palandri F, Martino B, Niederwieser D, Reiter A, Scott BL, Baer MR, Hoffman R, Odenike O, Vannucchi AM, Bussolari J, Zhu E, Rose E, Sherman L, Dougherty S, Sun L, Huang F, Wan Y, Feller FM, Rizo A, Kiladjian JJ. Randomized, Single-Blind, Multicenter Phase II Study of Two Doses of Imetelstat in Relapsed or Refractory Myelofibrosis. J Clin Oncol. 2021 Sep 10;39(26):2881-2892. doi: 10.1200/JCO.20.02864. Epub 2021 Jun 17. PMID 34138638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 55 investigative sites in Belgium, Canada, France, Germany, Israel, Italy, Korea, Spain, Taiwan, United Kingdom, and the United States from August 28, 2015, to 25 October 2016. Data analyses include all data through the data cut-off date February 07, 2020.
Pre-assignment Details: A total of 107 participants with Intermediate-2 or High-Risk Myelofibrosis (MF) Relapsed/Refractory to Janus Kinase (JAK) Inhibitor were randomly assigned to 1 of 2 treatment arms into 1:1 ratio to imetelstat 4.7 or imetelstat 9.4 mg/kg of body weight. Eligible participants were stratified based on a) spleen size ≥ 15 cm below the left costal margin by palpation (yes vs. no) and b) platelet count at study entry (platelets ≥75 x 10^9/L [Per Liter] and <150 x 10^9L vs. ≥150 x 10^9L).
Groups:
- Imetelstat 4.7 mg/kg: Participants received imetelstat 4.7 mg/kg of body weight as intravenous infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or study end. After the first interim analysis, treatment for all participants was unblinded and participants assigned to the imetelstat 4.7 mg/kg arm could continue with their same imetelstat dose or have it increased to 9.4 mg/kg at the investigator's discretion. After the end of main study, participants who were receiving benefit from study treatment opted to continue to receive imetelstat during the Extension Phase until there is loss of benefit or unacceptable toxicity. (Maximum duration on study was approximately 2.3 years and Maximum duration on extension phase was approximately 1.8 years).
- Imetelstat 9.4 mg/kg: Participants received imetelstat 9.4 mg/kg of body weight as intravenous infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or study end. After the end of the main study, participants who were receiving benefit from study treatment opted to continue to receive imetelstat during the Extension Phase until there is loss of benefit or unacceptable toxicity. (Maximum duration on study was approximately 2.3 years and Maximum duration on extension phase was approximately 1.8 years).
Period: Overall Study
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Started | 48 | 59
Treated | 48 | 59
Completed (Disposition data is reported until the end of study.) | 0 | 0
Not Completed | 48 | 59
Not completed — Death | 33 | 36
Not completed — Lost to Follow-up | 2 | 0
Not completed — Study Terminated by Sponsor | 5 | 14
Not completed — Withdrawal by Subject | 8 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis set included all participants randomized into the study and classified according to their assigned treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg | Total
Number analyzed (Participants) | 48 | 59 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.95) | 66.5 (9.39) | 67.2 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 40
  Male | 32 | 35 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 41 | 44 | 85
  Unknown | 2 | 3 | 5
  Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 48 | 88
  Black/African American | 2 | 2 | 4
  Asian | 2 | 3 | 5
  Multiple | 1 | 0 | 1
  Not Reported | 3 | 6 | 9
Region [Count of Participants; unit: Participants]
  United States/Canada | 25 | 18 | 43
  European Union | 19 | 34 | 53
  Rest of World | 4 | 7 | 11
Spleen Size by Palpation [Mean (Standard Deviation); unit: centimeter (cm)] — Population: Number analyzed signifies the number of participants with data available for spleen size palpitation.
  centimeter (cm)
    number analyzed (Participants) | 47 | 59 | 106
    (all) | 17.6 (7.62) | 17.3 (7.51) | 17.4 (7.53)
Platelet Count [Count of Participants; unit: Participants]
  <75 (10^9/L) | 1 | 2 | 3
  75 - <150 (10^9/L) | 23 | 31 | 54
  ≥150 (10^9/L) | 24 | 26 | 50
Eastern Cooperative Oncology Group (ECOG) Score [Count of Participants; unit: Participants] — ECOG Performance Score has 5 grades.0= Fully active, able to carry on all predisease performance without restriction;1= Restricted in physically strenuous activity but ambulatory and able to carry out work on a light or sedentary nature, eg, light housework, office work;2= Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours;3= Capable of only limited self-care; confined to bed or chair more than 50% of waking hours;4= Completely disabled. Cannot carry on any self-care.Totally confined to bed or chair;5= Dead.
  Participants
    0: Asymptomatic | 11 | 14 | 25
    1: Symptomatic fully ambulatory | 26 | 34 | 60
    2: Self care | 11 | 11 | 22
Time from Last JAKi Treatment [Median (Full Range); unit: months] | 1.4 [1 to 31] | 1.7 [1 to 38] | 1.7 [1 to 38]
Duration of Prior JAKi Treatment [Median (Full Range); unit: months] | 22.3 [3 to 90] | 24.5 [1 to 73] | 23.0 [1 to 90]
Dynamic International Prognostic Scoring System (DIPSS) [Count of Participants; unit: Participants] — DIPSS stratifies primary myelofibrosis (PMF) into four risk categories (low, intermediate 1, intermediate 2, and high risk), based on 5 clinical factors; Age>65, Hemoglobin <10gm/dL, Leukocytes >10 (9)/L, circulating blasts ≥1%, and constitutional symptoms.
  Participants
    Intermediate 2 | 28 | 34 | 62
    High Risk | 19 | 25 | 44
    Missing | 1 | 0 | 1
Type of Myelofibrosis (MF) [Count of Participants; unit: Participants]
  Primary MF (PMF) | 27 | 36 | 63
  Post Essential Thrombocythemia (PET) | 9 | 10 | 19
  Post Polycythemia Vera (PPV) | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Spleen Response
Description: Spleen response rate is defined as the percentage of participants who achieved ≥ 35% reduction in spleen volume at Week 24 from baseline performed by the IRC using magnetic resonance imaging (MRI).
Time Frame: Week 24
Population: Treated analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants | 0 [0 to 7.4] | 10.2 [3.8 to 20.8]

2. Primary Outcome: Percentage of Participants With Symptom Response
Description: Symptom response rate is defined as percentage of participants who achieved ≥ 50% reduction in total symptom score (TSS) at Week 24 from baseline as measured by the modified Myelofibrosis Symptom Assessment Form (MFSAF) version 2.0 diary. The MFSAF assessed following symptoms due to Myelofibrosis (MF): night sweats, itchiness, abdominal discomfort, pain under ribs on left side, feeling of fullness, bone or muscle pain and degree of inactivity. Each item is scored on a scale of 0 (absent) to 10 (worst imaginable) with higher scores indicating more severe symptoms and greater inactivity. The total score ranges from 0-70, where 0 indicates absent/as good as it can be and 70 indicates worst imaginable/as bad as it can be.
Time Frame: Week 24
Population: Treated analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants | 6.3 [1.3 to 17.2] | 32.2 [20.6 to 45.6]

3. Secondary Outcome: Percentage of Participants With Overall Response as Per Modified 2013 International Working Group - Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Criteria
Description: Overall Response Rate: % of participants with complete remission (CR) or partial remission (PR) per modified IWG-MRT.CR: bone marrow: normocellular <5% blasts, ≤Grade 1 fibrosis; immature myeloid cells in peripheral blood (PB):<2%;hemoglobin (Hb):10 g/dL-upper limit of normal (ULN); neutrophils:1*10^9/L-ULN; platelets: 100*10^9/L-ULN; spleen:not palpable and ≤350ml volume; extramedullary hematopoiesis (EMH): no non-hepato-splenic EMH; symptoms: >70% improvement in symptom score per modified MFSAF v2.0 TSS. PR: bone marrow: normocellular: <5% blasts ≤ Grade 1 fibrosis or not meeting bone marrow remission criteria; Immature myeloid cells in PB: <2%; Hb: 8.5 -<10 g/dL-ULN or 10 g/dL-ULN; neutrophils: 1*10^9/L-ULN; platelets: 50 -<100*10^9/L-ULN; spleen: ≥35% splenic volumetric reduction by MRI or not palpable; EMH: no non-hepato-splenic EMH;symptoms: >50% improvement in symptom score per modified MFSAF v2.0 TSS. All response categories, benefit must last >12 weeks to qualify as response.
Time Frame: Every 12 weeks up to Week 48 then every 24 weeks (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants | 0 [NA to NA] — Upper and lower limits of 95% CI was not estimable due to limited number of participants with the event. | 1.7 [0.0 to 9.1]

4. Secondary Outcome: Percentage of Participants With Clinical Improvement (CI) Per Modified 2013 IWG-MRT Criteria
Description: CI per the modified 2013 IWG-MRT criteria defined as the achievement of anemia, spleen or symptoms response without progressive disease or increase in severity of anemia, thrombocytopenia, or neutropenia (Increase in severity of anemia constitutes the occurrence of new transfusion dependency or a ≥ 2.0 g/dL decrease in hemoglobin level from pretreatment baseline that lasts for at least 12 weeks. Increase in severity of thrombocytopenia or neutropenia is defined as a 2-grade decline, from pretreatment baseline, in platelet count or ANC, according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. In addition, assignment to CI requires a minimum platelet count of ≥ 25,000*10^9/L and ANC of ≥ 0.5*10^9/L.) For all response categories, benefit must last for >12 weeks to qualify as a response.
Time Frame: Every 12 weeks up to Week 48 then every 24 weeks (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants | 16.7 | 25.4

5. Secondary Outcome: Percentage of Participants With Clinical Response Per Modified 2013 IWG-MRT
Description: Clinical response rate (CRR) was defined as percentage of participants who achieved CR, PR, or CI per modified 2013 IWG-MRT criteria. CR: bone marrow: normocellular <5% blasts, ≤Grade 1 fibrosis; immature myeloid cells in PB: <2%; Hb: 10 g/dL-ULN; neutrophils: 1*10^9/L-ULN; platelets: 100*10^9/L-ULN; spleen: not palpable and ≤350ml volume; EMH: no non-hepato-splenic EMH; symptoms: >70% improvement in symptom score per modified MFSAF v2.0 TSS. PR: bone marrow: normocellular: <5% blasts ≤ Grade 1 fibrosis or not meeting bone marrow remission criteria; Immature myeloid cells in PB: <2%; Hb: 8.5 -<10 g/dL-ULN or 10 g/dL-ULN; neutrophils: 1*10^9/L-ULN; platelets: 50 -<100*10^9/L-ULN; spleen: ≥35% splenic volumetric reduction by MRI or not palpable; EMH: no non-hepato-splenic EMH; symptoms: >50% improvement in symptom score per modified MFSAF v2.0 TSS. CI: achievement of anemia, spleen or symptoms response without PD or increase in severity of anemia, thrombocytopenia, or neutropenia.
Time Frame: Every 12 weeks up to Week 48 then every 24 weeks (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants | 16.7 [7.5 to 30.2] | 27.1 [16.4 to 40.3]

6. Secondary Outcome: Percentage of Participants With Spleen Response Per Modified 2013 IWG-MRT Criteria
Description: Spleen response per modified 2013 IWG-MRT criteria. Spleen response: a baseline splenomegaly that is palpable at 5-10 cm, below the left costal margin (LCM), becomes not palpable or a baseline splenomegaly that is palpable at >10 cm, below the LCM, decreases by ≥50%; A spleen response requires confirmation by MRI showing >35% spleen volume reduction (SVR). For response categories, benefit must last for >12 weeks to qualify as a response. Participants who achieved CI per modified IWG-MRT criteria considered as response with clinical improvement. Participants who met criteria for spleen response but had worsening cytopenias (and therefore did not meet criteria for clinical improvement) were considered to have a response without clinical improvement. The clinical improvement in IWG-MRT is defined as the achievement of anemia, spleen or symptoms response without progressive disease or increase in severity of anemia, thrombocytopenia, or neutropenia.
Time Frame: Every 12 weeks up to Week 48 then every 24 weeks (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug. All treated participants were evaluated for each response.
Measure: Number; unit: percentage of participants
Groups:
- Imetelstat 4.7 mg/kg: Participants received imetelstat 4.7 mg/kg of body weight as intravenous infusion on Day 1 of each cycle (each cycle was of 21 days) until disease progression, unacceptable toxicity, or study end. Participants had an option to continue the treatment at the current dose or escalated dose of 9.4 mg/kg based on investigator's discretion. After the end of main study, Participants who were receiving benefit from study treatment opted to continue to receive imetelstat during the Extension Phase until there is loss of benefit or unacceptable toxicity. (Maximum duration on study was approximately 2.3 years and Maximum duration on extension phase was approximately 1.8 years).
- Imetelstat 9.4 mg/kg: Participants received imetelstat 9.4 mg/kg of body weight as intravenous infusion on Day 1 of each cycle (each cycle was of 21 days) until disease progression, unacceptable toxicity, or study end. After the end of the main study, Participants who were receiving benefit from study treatment opted to continue to receive imetelstat during the Extension Phase until there is loss of benefit or unacceptable toxicity. (Maximum duration on study was approximately 2.3 years and Maximum duration on extension phase was approximately 1.8 years).
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants
  Spleen response with CI | 0 | 3.4
  Spleen response without CI | 2.1 | 0

7. Secondary Outcome: Percentage of Participants With Symptoms Response Per Modified 2013 IWG-MRT Criteria
Description: Symptoms response per modified 2013 IWG-MRT criteria. Symptoms Response: a ≥50% reduction in the modified MFSAF v2.0 TSS. For response category, benefit must last for >12 weeks to qualify as a response. Participants who achieved CI per modified IWG-MRT criteria considered as response with clinical improvement. Participants who met criteria for symptom response but had worsening cytopenias (and therefore did not meet criteria for clinical improvement) were considered to have a response without clinical improvement. The clinical improvement in IWG-MRT is defined as the achievement of anemia, spleen or symptoms response without progressive disease or increase in severity of anemia, thrombocytopenia, or neutropenia.
Time Frame: Every 12 weeks up to Week 48 then every 24 weeks (approximately up to 2.3 years)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants
  Symptom response with CI | 14.6 | 22.0
  Symptom response without CI | 4.2 | 8.5

8. Secondary Outcome: Percentage of Participants With Anemia Response Per Modified 2013 IWG-MRT Criteria
Description: Anemia response per modified 2013 IWG-MRT criteria. Anemia response is defined as participants with baseline Hb <10 g/dL but not meeting strict criteria for transfusion dependency: a ≥ 2 g/dL increase in Hb; Transfusion dependent participants at baseline: becoming transfusion independent. Transfusion independence is defined as absence of any pRBC transfusions for at least 12 "rolling" weeks. For response categories, benefit must last for >12 weeks to qualify as a response. Participants who achieved CI per modified IWG-MRT criteria considered as response with clinical improvement. Participants who met criteria for anemia response but had worsening cytopenias (and therefore did not meet criteria for clinical improvement) were considered to have a response without clinical improvement. The clinical improvement in IWG-MRT is defined as the achievement of anemia, spleen or symptoms response without progressive disease or increase in severity of anemia, thrombocytopenia, or neutropenia.
Time Frame: Every 12 weeks up to Week 48 then every 24 weeks (approximately up to 2.3 years)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
percentage of participants
  Anemia response with CI | 4.2 | 6.8
  Anemia response without CI | 0 | 1.7

9. Secondary Outcome: Duration of Response (PR/CI/RWCI) as Per IWG-MRT Criteria
Description: Duration of response (PR/CI/RWCI) is the duration from the date of initial documentation of a response to date of first documented evidence of PD or death, whichever occurs first. PR: BM: normocellular: <5% blasts ≤Grade 1 fibrosis/not meeting BM remission criteria; IMC in PB: <2%; Hb: 8.5 -<10 g/dL-ULN or 10 g/dL- ULN; neutrophils: 1*10^9/L-ULN; platelets: 50 -<100*10^9/L-ULN; spleen: ≥35% splenic volumetric reduction by MRI/not palpable; EMH: no non-hepato-splenic EMH; symptoms: >50% improvement in symptom score. CI: achievement of anemia, spleen or symptoms response without PD or increase in severity of anemia, thrombocytopenia, neutropenia. RWCI: Participants who met criteria for response but had worsening cytopenias. PD: Splenomegaly requires MRI showing ≥25% increase in spleen volume.
Time Frame: From date of initial documentation of a response to the date of first documented evidence of PD or death, whichever occurs first (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug. Here, "overall number of participants analyzed" signifies participants who were responders (PR/CI/RWCI) at any time.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 21
weeks | 36.3 [11.9 to 60.0] | 38.3 [27.0 to 48.3]

10. Secondary Outcome: Overall Survival
Description: Overall Survival is measured from the date of Cycle 1, Day 1 to the date of the participants death. If the participant's was alive or the vital status was unknown, OS was censored at the date that the participant is last known to be alive.
Time Frame: Day 1 of Cycle 1 (each cycle was of 21 days), up to the date of the participant's death (approximately up to 4.1 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
months | 19.91 [17.05 to 33.87] | 28.09 [22.80 to 31.61]

11. Secondary Outcome: Percentage of Participants With Clinically Meaningful Improvement in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-30 (QLQ-C30): Global Health Status
Description: EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients. The EORTC QLQ-C30 included 30 items resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) which are based on 4-point scale (1= Not at all to 4= Very much); and 1 global health status scale based on 7-point scale (1= Very poor to 7= Excellent). All scales and items are averaged, transformed to 0-100 scale; higher score=better level of functioning. Clinically meaningful improvement defined as change greater than half of the standard deviation at baseline in QLQ-C30 Global Health Status.
Time Frame: Up to end of the treatment (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug. Here, "overall number of participants analyzed" signifies the number of participants who had data at both baseline and end of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 18 | 33
percentage of participants | 22.2 | 36.4

12. Secondary Outcome: EuroQol 5 Dimension 5 Level (EQ-5D-5L): Utility Score and Visual Analog Scale (VAS)
Description: EQ-5D-5L is a standardized health-related quality of life questionnaire developed by EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L consists of two components: a health state profile and VAS. EQ-5D health state profile comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state. EQ-5D-5L- VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: At the end of treatment, up to approximately 2.3 years
Population: Treated analysis set included all participants who received at least 1 dose of study drug. Here "N"= participants who had data at both baseline and end of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 18 | 33
score on a scale
  EQ-5D-5L: Utility Score: number analyzed (Participants) | 18 | 32
  EQ-5D-5L: Utility Score | 0.498 (0.2999) | 0.626 (0.2117)
  EQ-5D-5L: VAS | 51.28 (21.143) | 47.73 (16.398)

13. Secondary Outcome: Percentage of Participants With Clinically Meaningful Improvement in Brief Pain Inventory (BPI)
Description: The BPI rates the intensity of pain on 4 items (right now, worst, least, and average), and the interference in 7 areas (general activity, mood, walking ability, normal work, relations, sleep, enjoyment of life). Minimum value = 0; maximum value = 10. Higher scores indicate greater symptom severity/worse outcomes. Clinically meaningful improvement in BPI defined as change greater than half of the standard deviation at baseline.
Time Frame: Up to end of treatment (approximately up to 2.3 years)
Population: Treated analysis set included all participants who received at least 1 dose of study drug. Here, "overall number of participants analyzed" signifies participants who had data at both baseline and end of treatment and "Number analyzed" signifies the number of participants with data available for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 18 | 33
percentage of participants
  Pain at its Worst: Improvement | 50.0 | 75.8
  Pain at its Least: Improvement | 44.4 | 51.5
  Pain on the Average: Improvement | 55.6 | 66.7
  Pain Right Now: Improvement | 61.1 | 66.7
  Relief Pain Treatments Provided: Improvement: number analyzed (Participants) | 18 | 32
  Relief Pain Treatments Provided: Improvement | 50.0 | 53.1
  Pain Interfered General Activity: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered General Activity: Improvement | 72.2 | 68.8
  Pain Interfered with Mood: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered with Mood: Improvement | 50.0 | 59.4
  Pain Interfered Walking Ability: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered Walking Ability: Improvement | 38.9 | 78.1
  Pain Interfered with Normal Work: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered with Normal Work: Improvement | 61.1 | 62.5
  Pain Interfered with Relations: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered with Relations: Improvement | 44.4 | 53.1
  Pain Interfered with Sleep: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered with Sleep: Improvement | 61.1 | 78.1
  Pain Interfered Enjoyment of Life: Improvement: number analyzed (Participants) | 18 | 32
  Pain Interfered Enjoyment of Life: Improvement | 61.1 | 62.5

14. Secondary Outcome: Patient's Global Impression of Change (PGIC)
Description: The PGIC was used to capture the participant's perspective of improvement or decline in MF symptoms over time. The PGIC had a 7-point response scale ranging from 1 to 7 where, (1=very much improved, 2= somewhat improved, 3= a little improved, 4=no change, 5= a little worse, 6= somewhat worse, 7=very much worse).
Time Frame: At the end of treatment, up to approximately 2.3 years
Population: Treated analysis set included all participants who received at least 1 dose of study drug. Here, "overall number of participants analyzed" signifies number of subjects who had data at both baseline and end of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 17 | 33
score on a scale | 4.82 (1.237) | 3.97 (1.571)

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were AEs with onset during or after the first dose of study drug, and within 30 days following the last dose of study drug.
Time Frame: Up to end of extension phase (approximately up to 4.2 years)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 48 | 59
Participants | 47 | 59

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Imetelstat
Time Frame: 0 (before start of infusion), 1, 2, 3-5, 6-10, 12-16 and 18-24 hours post dose on Day 1 of Cycle 1 (each cycle was of 21 days)
Population: Pharmacokinetic (PK) subset included all participants who had serial PK sampling during cycle 1 treatment to determine the maximum plasma concentration of Imetelstat by noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- PK: Imetelstat 4.7 mg/kg: Participants received imetelstat 4.7 mg/kg of body weight as intravenous infusion on Day 1 of cycle 1 and those who had serial PK samples collected.
- PK: Imetelstat 9.4 mg/kg: Participants received imetelstat 9.4 mg/kg of body weight as intravenous infusion on Day 1 of cycle 1 and those who had serial PK samples collected.
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
μg/mL | 57.0 (72.3) | 81.9 (40.0)

17. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Imetelstat
Time Frame: as for outcome 16
Population: PK subset included all participants who had serial PK sampling during cycle 1 treatment to determine the time to reach maximum plasma concentration of imetelstat by noncompartmental PK analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
hr | 2.00 [1.93 to 2.20] | 2.00 [1.00 to 2.75]

18. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC 0-24) of Imetelstat
Time Frame: as for outcome 16
Population: PK subset included all participants who had serial PK sampling during cycle 1 treatment to determine the AUC 0-24 of Imetelstat by noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
μg*hr/mL | 171 (135) | 501 (283)

19. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Infinity (AUC0-inf) of Imetelstat
Time Frame: as for outcome 16
Population: PK subset included all participants who had serial PK sampling during cycle 1 treatment to determine AUC 0-inf of Imetelstat by noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
μg*h/mL | 193 (156) | 524 (297)

20. Secondary Outcome: Elimination Half-Life (t1/2) of Imetelstat
Description: Elimination half-life (t 1/2) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Time Frame: as for outcome 16
Population: PK subset included all participants who had serial PK sampling during cycle 1 treatment to determine the t1/2 of Imetelstat by noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
hr | 4.6 (1.6) | 5.5 (1.5)

21. Secondary Outcome: Total Systemic Clearance (CL) of Imetelstat
Time Frame: as for outcome 16
Population: PK subset included all participants who had serial PK sampling during cycle 1 treatment to determine the CL of Imetelstat by noncompartmental PK analysis.
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
L/hr/kg | 0.0329 (0.0138) | 0.0252 (0.0157)

22. Secondary Outcome: Volume of Distribution (Vd) of Imetelstat
Time Frame: as for outcome 16
Population: PK population analysis set included all participants who received at least 1 dose of study drug and had at least 1 sample collected during treatment to determine the drug concentration.
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | PK: Imetelstat 4.7 mg/kg | PK: Imetelstat 9.4 mg/kg
Number analyzed (Participants) | 11 | 17
L/kg | 0.198 (0.0770) | 0.190 (0.104)

ADVERSE EVENTS:
Time Frame: Up to end of extension phase (approximately up to 4.2 years)
Description: Safety analysis set included all participants who received at least 1 dose of study treatment.
Groups:
- Imetelstat 4.7 mg/kg: Participants received imetelstat 4.7 mg/kg of body weight as intravenous infusion on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or study end. After the first interim analysis, treatment for all participants was unblinded and participants assigned to the imetelstat 4.7 mg/kg arm could continue with their same imetelstat dose. After the end of main study, participants who were receiving benefit from study treatment opted to continue to receive imetelstat during the Extension Phase until there is loss of benefit or unacceptable toxicity. (Maximum duration on study was approximately 2.3 years and Maximum duration on extension phase was approximately 1.8 years). AEs for the 12 subjects whose dose was later escalated are included here for the period before dose escalation.
- Imetelstat Dose Escalated From 4.7 mg/kg to 9.4 mg/kg: Participants initially treated with 4.7 mg/kg imetelstat in Imetelstat 4.7 mg/kg arm group were subsequently dose escalated to 9.4 mg/kg at the investigator's discretion. Dose escalation for these participants may occur at any cycle (each of 21-day cycle) of the treatment phase. After the end of main study, participants who were receiving benefit from study treatment opted to continue to receive imetelstat during the Extension Phase until there is loss of benefit or unacceptable toxicity. (Maximum duration on study was approximately 2.3 years and Maximum duration on extension phase was approximately 1.8 years). AEs reported in this column occurred after dose escalation.
Arm/Group | Imetelstat 4.7 mg/kg | Imetelstat 9.4 mg/kg | Imetelstat Dose Escalated From 4.7 mg/kg to 9.4 mg/kg
All-Cause Mortality (participants affected / at risk) | 34/48 | 36/59 | 1/12
Serious Adverse Events (participants affected / at risk) | 24/48 | 21/59 | 4/12
Other Adverse Events (participants affected / at risk) | 47/48 | 59/59 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imetelstat 4.7 mg/kg (N=48) | Imetelstat 9.4 mg/kg (N=59) | Imetelstat Dose Escalated From 4.7 mg/kg to 9.4 mg/kg (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Splenic artery thrombosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 2 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imetelstat 4.7 mg/kg (N=48) | Imetelstat 9.4 mg/kg (N=59) | Imetelstat Dose Escalated From 4.7 mg/kg to 9.4 mg/kg (N=12)
Anaemia (Blood and lymphatic system disorders) | 15 | 26 | 5
Leukocytosis (Blood and lymphatic system disorders) | 3 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 8 | 2
Neutropenia (Blood and lymphatic system disorders) | 5 | 21 | 3
Splenomegaly (Blood and lymphatic system disorders) | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 29 | 4
Palpitations (Cardiac disorders) | 2 | 6 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 14 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0
Constipation (Gastrointestinal disorders) | 9 | 9 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 18 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 15 | 20 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 9 | 8 | 1
Asthenia (General disorders) | 9 | 14 | 1
Chills (General disorders) | 3 | 8 | 0
Fatigue (General disorders) | 10 | 15 | 1
Malaise (General disorders) | 2 | 3 | 0
Oedema peripheral (General disorders) | 13 | 10 | 3
Pain (General disorders) | 1 | 3 | 0
Pyrexia (General disorders) | 8 | 13 | 2
Nasopharyngitis (Infections and infestations) | 0 | 6 | 0
Rhinovirus infection (Infections and infestations) | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 9 | 1
Urinary tract infection (Infections and infestations) | 2 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 5 | 0
Serum ferritin increased (Investigations) | 0 | 4 | 0
Weight decreased (Investigations) | 9 | 8 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 10 | 1
Gout (Metabolism and nutrition disorders) | 2 | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1
Dizziness (Nervous system disorders) | 2 | 10 | 1
Headache (Nervous system disorders) | 6 | 10 | 1
Insomnia (Psychiatric disorders) | 6 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 15 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 8 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 6 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 1
Hypertension (Vascular disorders) | 3 | 4 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 2
Genital ulceration (Reproductive system and breast disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hot flush (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consistent with Good Publication Practices and ICMJE guidelines, the sponsor shall have right to publish such primary (multicenter) data and information without approval from investigator. Investigator has right to publish study site-specific data after primary data published. If an investigator wishes to publish information from study, a copy of manuscript must be provided to sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02426086/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT02426086/SAP_001.pdf